CLINICAL TRIAL: NCT04917575
Title: Efficacy Trial of Life Simulation Game to Routinize Adolescent HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Media Rez (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCR191708
Record Dates: First submitted 2021-05-20; First posted 2021-06-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hiv
Keywords: HIV prevention; HIV testing; mHealth; Pre-exposure prophylaxis (PrEP); adolescents; interactive technology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Game (Experimental): An enhanced life-simulation prototype of a playable interactive game to increase HIV testing, risk assessment tool, and HIV and pre-exposure prophylaxis (PrEP) locators embedded within the game.
  Interventions: Other: Mobile Game
- Mobile Application (Active Comparator): A mobile application that will include basic information on HIV basics (e.g., routes of transmission, data on the epidemiology of HIV among youth), prevention information on HIV testing and PrEP, as well as a link to the HIV risk estimator, and HIV testing and PrEP locators.
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Game — An enhanced life-simulation prototype of a playable interactive game to increase HIV testing.
  Arms: Mobile Game
Other: Mobile Application — A mobile application that will include basic information on HIV basics (e.g., routes of transmission, data on the epidemiology of HIV among youth), prevention information, and information on HIV testing and PrEP, as well as a link to the HIV risk estimator, and HIV testing and PrEP locators.
  Arms: Mobile Application

SUMMARY:
This study will aim to assess the acceptability, usability and efficacy of using state-of-the-art video game technology to increase HIV testing among adolescents and young adults (AYA) ages 13-24. AYA often lack awareness of their personal risk of contracting HIV and where to go for testing and care. This lack of awareness has contributed to poor uptake of HIV testing among AYA despite engagement in high risk behaviors. The goal of this project is to harness this strong motivation to play games to increase HIV testing. Previous games for behavior change have yielded early success for increasing target behaviors among their sample populations, yet research on increasing HIV testing among AYA through gaming has been limited. This intervention builds on prior formative work and is designed to offer AYA personally-tailored risk messages and supports their accessibility to HIV testing and prevention services through an innovative gaming approach that is sharable over social media with in-game rewards for sharing the game with peers. The specific aim of this study is to determine the efficacy of a life-simulation game in changing HIV testing, knowledge, and risk behaviors among AYA at risk for HIV.

ELIGIBILITY:
Inclusion Criteria:

* age 13-24
* self-reported HIV negative or unknown status
* self-reported ever sexually active
* resident of the DC metropolitan region which includes the District of Columbia, Maryland and Virginia for at least the next 6 months
* Is able to provide informed consent or assent
* able to complete all study procedures in English
* has own mobile phones and be willing to use them for the study.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
HIV testing | prior 6 months
  Self-reported HIV testing in the past 6 months

SECONDARY OUTCOMES:
Intent to test for HIV | baseline, 1, 3, 6 months
  Intent to test will be assessed using a validated 6-point Likert scale
HIV knowledge | baseline, 1, 3, 6 months
  18-item scale
HIV risk perception and behaviors | baseline, 1, 3, 6 months
  8-item scale and perceived likelihood of getting infected (0-100%)
Knowledge of PrEP | baseline, 1, 3, 6 months
  Has participant heard of PrEP at specified time period
CDC risk estimator scores | baseline, 1, 3, 6 months
Frequency of game use | 1, 3, 6 months
PrEP screening | baseline, 1, 3, 6 months
  ever been screened for PrEP eligibility
PrEP use/uptake | baseline, 1, 3, 6 months
  been prescribed/taken PrEP
PrEP locator use | baseline, 1, 3, 6 months
  Number of linkages to PrEP locator
Duration of game use | 1, 3, 6 months
Reasons for continued or discontinued use of game | 1, 3, 6 months
HIV locator use | baseline, 1, 3, 6 months
  Number of linkage to HIV testing locator

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Milken School of Public Health, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Castel AD, Wilbourn B, Trexler C, D'Angelo LD, Greenberg D. A Digital Gaming Intervention to Improve HIV Testing for Adolescents and Young Adults: Protocol for Development and a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 24;10(6):e29792. doi: 10.2196/29792. PMID 34185022